CLINICAL TRIAL: NCT00038207
Title: Phase II Liposomal Vincristine for Pediatric and Adolescent Patients With Relapsed Malignancies
Brief Title: Liposomal Vincristine for Pediatric and Adolescent Patients With Relapsed Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Inex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P99-401
Record Dates: First submitted 2002-05-29; First posted 2002-05-30 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Soft Tissue Sarcoma; Lymphoma; Leukemia; Wilms' Tumor; Osteosarcoma
Keywords: soft tissue sarcoma; Bone sarcomas
MeSH Terms: conditions — Sarcoma; Lymphoma; Leukemia; Wilms Tumor; Osteosarcoma; Bone Neoplasms | interventions — Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liposomal Vincristine (Experimental)
  Interventions: Drug: Liposomal Vincristine

INTERVENTIONS:
Drug: Liposomal Vincristine — Vincristine Sulfate Liposome Injection (VSLI) administered via a central venous catheter at 2.0 mg/m2 over 60 minutes every 14 days + 2 days
  Other Names: Vincristine Sulfate Liposome

SUMMARY:
The goal of this clinical research study is to learn if treatment with the drug liposomal vincristine can shrink or slow the growth of the patient's cancer. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Before and during the treatment patients will have exams done. These may include blood tests, urine tests, bone marrow tests, tests of the central nervous system, x-rays, or MRI/CT test. These are needed to measure the patient's clinical condition and progress. A physical exam and blood tests (about 2 teaspoons) will be repeated at least one time weekly.

Since Liposomal Vincristine may prevent the body from making and/or keeping new blood cells, prior to treatment patients will also have a Human Immunodeficiency Virus (AIDS virus) test, a blood test to detect the presence of antibodies to the AIDS virus. A separate informed consent will be given to be signed, in order to obtain permission for this test. Female patients may also be required to have a urine pregnancy test before treatment may begin, as it is not known how the drug may affect the unborn child.

Patients will receive liposomal vincristine through a central venous catheter (a plastic tube usually inserted under the collar bone) over one hour, once every 14 days, + 2 days. Patient's will also be given the drug docusate by the day liposomal vincristine is started. This is done to try to prevent constipation as a side effect.

All patients who show a continued response or stable disease without major side effects may continue to receive liposomal vincristine for up to 24 months. Patients with solid tumors and lymphoma will have X-rays performed every 8 weeks to follow the progression of their tumor. Patients with leukemia will have a bone marrow aspirate and biopsy done after the first and second months of treatment, and then every 8 weeks.

This is an investigational study. The FDA has authorized the use of the study drug in research. Up to 60 patients will take part in this study. Up to 30 patients will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed malignancies in the following strata: (As of 09/01/02, the soft tissue sarcoma strata will remain open for new patient accrual. Strata listed in b, c, d, e will be closed to entry).

  1. soft tissue sarcoma
  2. bone sarcoma(CLOSED TO ENTRY AS OF 09/01/02)
  3. Wilms tumor(CLOSED TO ENTRY AS OF 09/01/02)
  4. lymphoma(CLOSED TO ENTRY AS OF 09/01/02)
  5. leukemia(CLOSED TO ENTRY AS OF 09/01/02)
* Performance status: Zubrod less than 3. Patients with long standing limited mobility requiring the use of a wheelchair will be considered ambulatory for the purpose of this protocol.
* Bidimensionally measurable disease radiologically.
* No anti-cancer treatment within the past 3 weeks.
* ANC greater than or equal to 500; platelets greater than or equal to 50,000; bilirubin less than or equal to 1.5 mg/dl; SGPT less than or equal to 4 x upper normal limit; creatinine less than or equal to 2 x normal. Patients with bone marrow infiltrative disease may be entered irrespective of ANC or platelets.
* Patients may be enrolled after BMT or PSCT if they meet all the above eligibility criteria.

Exclusion criteria:

* HIV positive.
* Serious intercurrent illness, active infections, or second cancer except basal cell carcinoma of the skin or cervical carcinoma in situ.
* Eligible for treatment of a higher priority.
* Pregnancy.
* Grade 3 or 4 sensory or motor dysfunction due to prior vinca alkaloids.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2000-06; Primary Completion 2004-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Response | 3 Months post initiation of treatment
  Response defined as Complete Response or Partial Response.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia E. Herzog, MD, BA, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org